CLINICAL TRIAL: NCT03398889
Title: Intestinal Microbiome and Extremes of Atherosclerosis
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 105166
Record Dates: First submitted 2017-12-12; First posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Gastrointestinal Microbiome, Atherosclerosis, Nutrients; Renal Function
Keywords: intestinal microbiome; atherosclerosis; nutrients; renal function
MeSH Terms: conditions — Atherosclerosis | interventions — Gastrointestinal Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA samples stored
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Unexplained Atherosclerosis phenotype: Residual score in linear regression >2
  Interventions: Diagnostic Test: Plasma levels of metabolites; Behavioral: Dietary questionnaire; Diagnostic Test: Intestinal microbiome
- Explained Atherosclerosis phenotype: Residual score in linear regression <-2, <2
  Interventions: Diagnostic Test: Plasma levels of metabolites; Behavioral: Dietary questionnaire; Diagnostic Test: Intestinal microbiome
- Protected Atherosclerosis phenotype: Residual score <-2
  Interventions: Diagnostic Test: Plasma levels of metabolites; Behavioral: Dietary questionnaire; Diagnostic Test: Intestinal microbiome

INTERVENTIONS:
Diagnostic Test: Plasma levels of metabolites — plasma levels of metabolites
Behavioral: Dietary questionnaire — Harvard food frequency questionnaire
Diagnostic Test: Intestinal microbiome — amplification and sequencing of 16S rRNA gene variable regions in stool samples

SUMMARY:
Patients attending stroke prevention clinics and a premature atherosclerosis clinic at University Hospital in London, ON, Canada were recruited to the study. They completed a dietary questionnaire, provided stool samples and had blood drawn to measure plasma levels of metabolites produced by the intestinal bacteria.

DETAILED DESCRIPTION:
Patients were phenotyped by their residual score in linear multiple regression with measured carotid plaque burden as the dependent variable and coronary risk factors were predictors. The residual score essentially represents the distance off the regression line of predicted plaque. They were grouped into three categories: Unexplained atherosclerosis (with more plaque than predicted by risk factors; residual score >2); Explained (the amount of plaque predicted by risk factors, residual score >-2 and <2); and Protected (less plaque than predicted by risk factors, residual score <-2).

DNA was extracted from stool samples in the lab of Dr. Allen-Vercoe at University of Guelph. RNA makeup of the intestinal microbiome was assessed in the lab of Dr. Gregory Gloor at Western. Plasma levels of trimethylamine n-oxide, p-cresylsulfate, hippuric acid, p-cresyl glucuronide, pheny acetyl glutamine and phenyl sulfate were measured by ultra-performance liquid chromatography coupled to quadrupole time-of-flight mass spectrometry in the lab of Dr. Bradley Urquhart at Western.

Nutrient intake over the past year was calculated at the Harvard School of Public Health from the 131 item self-reported and semi-quantitative Harvard Food Frequency Questionnaire (FFQ).

Estimated glomerular filtration rate was calculated from the Chronic Kidney Disease Epidemiological (CKD-EPI) equations.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending stroke prevention clinics and a Premature Atherosclerosis Clinic at University Hospital, London, ON, Canada,
* with measurements of carotid plaque burden and the risk factors used in the linear regression model.
* Willing to consent to the protocol approved by the Ethics board

Exclusion Criteria:

* Missing data on variables used in the regression model,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male, female
Study Population: as above
Sampling Method: Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2016-10-15 (Actual); Study Completion 2016-10-15 (Actual)

PRIMARY OUTCOMES:
Plasma levels of metabolites in the three phenotypes | Day 1
  Plasma levels of trimethylamine n-oxide, p-cresylsulfate, hippuric acid, p-cresyl glucuronide, pheny acetyl glutamine and phenyl sulfate

SECONDARY OUTCOMES:
Bacterial profile of the intestinal microbiome | Day 1
  Amplification and sequencing of 16S rRNA gene variable regions
Effect of nutrient intake on plasma levels of metabolites | Day 1
  Nutrient analysis from food frequency questionnaire
Effect of renal function on plasma levels of metabolites | Day 1
  eGFR from CKD-EPI equations

CONTACTS AND LOCATIONS:
Locations (1):
- Stroke Prevention & Atherosclerosis Research Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
It will depend on requests.